CLINICAL TRIAL: NCT00494975
Title: The Effect of Phototherapy on Pruritus of Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200704019R
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2010-09

CONDITIONS: Uremic Pruritus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB-UVB (Experimental): Narrow band-Ultraviolet B phototherapy
  Interventions: Device: Narrow band UVB phototherapy , long wave UVA phototherapy
- UVA (Placebo Comparator): Ultraviolet A Phototherapy
  Interventions: Device: Narrow band UVB phototherapy , long wave UVA phototherapy

INTERVENTIONS:
Device: Narrow band UVB phototherapy , long wave UVA phototherapy — A UV irradiation cubicle (HOUVA II, National Biological Corporation, OH, U.S.A.) equipped with 24 UVA lamps (F72T12/BL9/HO UVA, National Biological Corporation, OH, U.S.A. ) and 24 UVB lamps (TL100W/01 311NB UVB, Philips Company, Eindhoven, The Netherlands).

SUMMARY:
The purpose of this study was to confirm the efficacy of NB UVB phototherapy in alleviating uremic pruritus and investigate the association between improvement of pruritus and change of serum parameters, including routine biochemical data, immune profile and dialysis adequacy.

DETAILED DESCRIPTION:
We would conduct a randomized study to evaluate the effect of NB UVB therapy on uremic pruritus. The intensity of pruritus will be evaluated using visual analog scale (VAS) score (0 [no pruritus]-10 most severe pruritus]) and a detailed questionnaire assessing various characteristics of pruritus at baseline . The patients with the intensity of pruritus VAS score more than 5 will be randomized to narrow band UVB and control group. Phototherapy was administered to the whole body surface 2-3 sessions per week for total 18 sessions in a UV irradiation cubicle. The dose increased from 210mJ/cm2 .Doses were increased by 10 % at every session. The control group received time-matched exposures to long-wave ultraviolet light. The investigator will determine the pruritic intensity at baseline every 3 sessions by VAS score and by detailed questionnaire at baseline and after 18 sessions. The blood sample will also be collected at baseline and after treatment to determine factors associated with improvement.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease with moderate to severe uremic pruritus for longer than 2 months

Exclusion Criteria:

* pregnancy history of photosensitivity photo-aggravated disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ju Ko, MD, Principal Investigator — Nationa l Taiwan University Hospital Yun-Lin branch
Locations (1):
- Department of dermatology, National Taiwan Univeristy Hospital Yun-Lin branch, Douliu, Yunlin County, Taiwan

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264
- [Derived] Ko MJ, Yang JY, Wu HY, Hu FC, Chen SI, Tsai PJ, Jee SH, Chiu HC. Narrowband ultraviolet B phototherapy for patients with refractory uraemic pruritus: a randomized controlled trial. Br J Dermatol. 2011 Sep;165(3):633-9. doi: 10.1111/j.1365-2133.2011.10448.x. PMID 21668425

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultraviolet A Phototherapy: a UV irradiation cubicle (HOUVA II, National Biological Corporation, OH, U.S.A.) equipped with 24 UVA lamps (F72T12/BL9/HO UVA, National Biological Corporation, OH, U.S.A. )
- Narrow Band Ultraviolet B Phototherapy: a UV irradiation cubicle (HOUVA II, National Biological Corporation, OH, U.S.A.) equipped with 24 UVB lamps (TL100W/01 311NB UVB, Philips Company, Eindhoven, The Netherlands).
Period: Overall Study
Arm/Group | Ultraviolet A Phototherapy | Narrow Band Ultraviolet B Phototherapy
Started | 10 | 11
Completed | 8 | 10
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultraviolet A Phototherapy | Narrow Band Ultraviolet B Phototherapy | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 5 | 4 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.3) | 60.9 (11.5) | 62.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Taiwan | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Score for Pruritus
Description: a VAS is a horizontal line, 100 mm in length. The patient marks on the line the point that they feel represents their perception of their pruritus.
  0 (no pruritus) - 10 (most severe pruritus) The investigator will determine the pruritic intensity at baseline, every 3 sessions by VAS score, and by detailed questionnaire at baseline and after 18 sessions
Time Frame: VAS score at baseline and after 6 -week phototherapy
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ultraviolet A Phototherapy | Narrow Band Ultraviolet B Phototherapy
Number analyzed (Participants) | 8 | 10
Units on a scale | -3.38 (2.59) | -3.53 (3.49)
Statistical Analysis 1: Comparison: Ultraviolet A Phototherapy vs Narrow Band Ultraviolet B Phototherapy; The VAS score of pruritus intensity was recorded for each participant at baseline and weekly until week 12 so that each one had 12 repeatedly measured data scores. To investigate the predictive effects of age, sex, comorbid diseases, phototherapy, and results of blood laboratory exams on the intensity of pruritus, marginal linear regression model was fitted to the repeatedly measured VAS score data using the generalized estimating equations (GEE) method; Test type: Superiority or Other; p < 0.05, generalized estimating equations (GEE); Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.31 to 1.56], Standard Error of Mean 0.32

2. Secondary Outcome: Detailed Questionnaire at Baseline and After 18 Sessions
Time Frame: at baseline and after 18 sessions
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Arm/Group | Ultraviolet A Phototherapy | Narrow Band Ultraviolet B Phototherapy
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes